CLINICAL TRIAL: NCT01253291
Title: An Open-Label Extension Study of Multiple Subcutaneous Doses of LY2127399 in Japanese Patients With Rheumatoid Arthritis Treated With Methotrexate
Brief Title: A Study of Japanese Rheumatoid Arthritis Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13417; H9B-JE-BCDL (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-12-01; First posted 2010-12-03 (Estimated); Results first posted 2019-03-01 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2018-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tabalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 30mg/120 mg LY2127399 (Experimental): Participants in the 30 milligrams (mg) every 4 weeks arm of the lead-in study will receive 30 mg every 4 weeks until the safety of the 120 mg every 4 weeks dose is confirmed in the lead-in study.
  Interventions: Drug: LY2127399
- 120 mg LY2127399 (Experimental): Participants in the 60 mg every 4 weeks, 120 mg every 4 weeks and 120 mg every 2 weeks arms of the lead-in study will receive 120 mg every 4 weeks as these participants will enroll in this study after the safety of the 120 mg every 4 weeks dose in the lead-in study is confirmed.
  Interventions: Drug: LY2127399

INTERVENTIONS:
Drug: LY2127399 — Administered subcutaneously every 4 weeks for 48 weeks
  Other Names: tabalumab

SUMMARY:
The objective of this study is to evaluate the safety and tolerability of 48 weeks subcutaneous (SC) dosing with LY2127399 for participants who have participated in a prior LY2127399 clinical study. At the end of the 48-week treatment period, participants will participate in a 24-week follow-up period. Additional follow up after Week 72 may continue to assess B-cell recovery.

ELIGIBILITY:
Inclusion criteria

* Have given written informed consent
* Women must not be pregnant, breastfeeding or be at risk to become pregnant during study participation
* Must have completed treatment and 12 week follow up period in prior LY2127399 study NCT01253226 [Study H9B-JE-BCDK (BCDK)]

Exclusion criteria

* Have had any safety event during the previous LY2127399 (BCDK) study that participants participated in
* Have received, during previous study (BCDK), any drugs prohibited in the study protocol which includes unapproved drugs, live vaccines, or any biologic or non-biologic disease-modifying anti-rheumatic drug (DMARD) except for, methotrexate (MTX), hydroxychloroquine, sulfasalazine or bucillamine

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-05; Primary Completion 2013-09 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY(1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM-5 PM Eastern time (UTC/GMT - 5 hours, EST ), Study Director — Eli Lilly and Company
Locations (9):
- Japan (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aichi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukui
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gunma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ibaraki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miyagi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who completed NCT01253226 [Study H9B-JE-BCDK (BCDK)] were enrolled into open-label study NCT01253291 [H9B-JE-BCDL (BCDL]).
Groups:
- Placebo/LY2127399 120 mg Q4W: Participants who previously received placebo in Study BCDK were assigned to receive 120 milligrams (mg) of LY2127399 administered subcutaneously (SC) once every 4 weeks (Q4W) for 48 weeks.
- LY2127399 30 mg Q4W/120 mg Q4W: Participants who previously received 30 mg of LY2127399 Q4W in Study BCDK were assigned to receive 120 mg of LY2127399 administered SC Q4W for 48 weeks.
- LY2127399 60 mg Q4W/120 mg Q4W: Participants who previously received 60 mg of LY2127399 Q4W in Study BCDK were assigned to receive 120 mg of LY2127399 administered SC Q4W for 48 weeks.
- LY2127399 120 mg Q4W/120 mg Q4W: Participants who previously received 120 mg of LY2127399 Q4W in Study BCDK were assigned to receive 120 mg of LY2127399 administered SC Q4W for 48 weeks.
- LY2127399 120 mg Q2W/120 mg Q4W: Participants who previously received 120 mg of LY2127399 every 2 weeks (Q2W) in Study BCDK were assigned to receive 120 mg of LY2127399 administered SC Q4W for 48 weeks.
Period: Overall Study
Arm/Group | Placebo/LY2127399 120 mg Q4W | LY2127399 30 mg Q4W/120 mg Q4W | LY2127399 60 mg Q4W/120 mg Q4W | LY2127399 120 mg Q4W/120 mg Q4W | LY2127399 120 mg Q2W/120 mg Q4W
Started | 6 | 6 | 4 | 5 | 5
Received Study Drug During BCDL | 6 | 6 | 4 | 5 | 5
Completed | 2 | 4 | 4 | 5 | 3
Not Completed | 4 | 2 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Placebo/LY2127399 120 mg Q4W: Participants who previously received placebo in Study BCDK were assigned to receive 120 mg of LY2127399 administered SC Q4W for 48 weeks.
- LY2127399 120 mg Q2W/120 mg Q4W: Participants who previously received 120 mg of LY2127399 Q2W in Study BCDK were assigned to receive 120 mg of LY2127399 administered SC Q4W for 48 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo/LY2127399 120 mg Q4W | LY2127399 30 mg Q4W/120 mg Q4W | LY2127399 60 mg Q4W/120 mg Q4W | LY2127399 120 mg Q4W/120 mg Q4W | LY2127399 120 mg Q2W/120 mg Q4W | Total
Number analyzed (Participants) | 6 | 6 | 4 | 5 | 5 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (17.4) | 66.5 (5.7) | 47.8 (16.9) | 53.8 (14.1) | 55.8 (8.6) | 56.4 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 2 | 3 | 4 | 20
  Male | 1 | 0 | 2 | 2 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 4 | 5 | 5 | 26
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 6 | 6 | 4 | 5 | 5 | 26
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 6 | 6 | 4 | 5 | 5 | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: Included are the number of participants who experienced SAEs and treatment-emergent other non-SAEs. A summary of SAEs and other non-SAEs, regardless of causality, is located in the Reported Adverse Events (AEs) module.
Time Frame: Baseline up to 72 weeks
Population: All enrolled participants who received at least 1 dose of study drug during BCDL.
Measure: Count of Participants; unit: Participants
Groups:
- LY2127399 30 mg Q4W/120 mg Q4W: Participants who previously received 30 mg Q4W of LY2127399 in Study BCDK were assigned to receive 120 mg of LY2127399 administered SC Q4W for 48 weeks.
- LY2127399 60 mg Q4W/120 mg Q4W: Participants who previously received 60 mg Q4W of LY2127399 in Study BCDK were assigned to receive 120 mg of LY2127399 administered SC Q4W for 48 weeks.
- LY2127399 120 mg Q4W/120 mg Q4W: Participants who previously received 120 mg Q4W of LY2127399 in Study BCDK were assigned to receive 120 mg of LY2127399 administered SC Q4W for 48 weeks.
- LY2127399 120 mg Q2W/120 mg Q4W: Participants who previously received 120 mg Q2W of LY2127399 in Study BCDK were assigned to receive 120 mg of LY2127399 administered SC Q4W for 48 weeks.
Arm/Group | Placebo/LY2127399 120 mg Q4W | LY2127399 30 mg Q4W/120 mg Q4W | LY2127399 60 mg Q4W/120 mg Q4W | LY2127399 120 mg Q4W/120 mg Q4W | LY2127399 120 mg Q2W/120 mg Q4W
Number analyzed (Participants) | 6 | 6 | 4 | 5 | 5
Participants
  SAEs | 0 | 0 | 0 | 0 | 0
  Treatment Emergent Other Non-Serious AEs | 5 | 4 | 4 | 3 | 4

2. Secondary Outcome: Percent Change From Baseline in Anti-Cyclic Citrullinated Peptide (Anti-CCP) Antibody
Description: Anti-CCP is a disease related peripheral blood biomarker used to assess disease progression of rheumatoid arthritis (RA). A reduction in anti-CCP values indicates an improvement.
Time Frame: Baseline and Weeks 12, 24, 36, 52, and 72
Population: All enrolled participants with an anti-CCP antibody assessment at 1 or more of the specified timepoints.
Measure: Mean (Standard Deviation); unit: Percent Change of Anti-CCP
Groups:
- 120 mg LY2127399 Q4W: Participants who previously received placebo or 30 mg Q4W up to 120 mg Q4W of LY2127399 in Study BCDK were assigned to receive 120 mg of LY2127399 administered SC Q4W for 48 weeks.
Arm/Group | 120 mg LY2127399 Q4W
Number analyzed (Participants) | 9
Percent Change of Anti-CCP
  Anti-CCP Week 12: number analyzed (Participants) | 7
  Anti-CCP Week 12 | 19.9 (54.4)
  Anti-CCP Week 24: number analyzed (Participants) | 7
  Anti-CCP Week 24 | 8.5 (43.8)
  Anti-CCP Week 36 | -1.2 (19.7)
  Anti-CCP Week 52: number analyzed (Participants) | 8
  Anti-CCP Week 52 | 17.4 (50.7)
  Anti-CCP Week 72: number analyzed (Participants) | 7
  Anti-CCP Week 72 | -4.4 (31.7)

3. Secondary Outcome: Percent Change From Baseline in Rheumatoid Factor (RF)
Description: RF is a disease-related, peripheral blood biomarker used to assess disease progression of RA. A reduction in RF values indicate an improvement in RA symptoms.
Time Frame: Baseline and Weeks 12, 24, 36, 52, and 72
Population: All enrolled participants who had 1 or more RF assessment at 1 or more of the specified timepoints.
Measure: Mean (Standard Deviation); unit: Percent Change of RF
Arm/Group | 120 mg LY2127399 Q4W
Number analyzed (Participants) | 20
Percent Change of RF
  RF Week 12 | -2.0 (67.0)
  RF Week 24: number analyzed (Participants) | 19
  RF Week 24 | -9.7 (47.8)
  RF Week 36: number analyzed (Participants) | 18
  RF Week 36 | -7.9 (57.3)
  RF Week 52: number analyzed (Participants) | 16
  RF Week 52 | -2.3 (63.7)
  RF Week 72: number analyzed (Participants) | 16
  RF Week 72 | 25.3 (98.0)

4. Secondary Outcome: Percent Change From Baseline in Immunoglobulins [Immunoglobulin (Ig) G, IgM, and IgA]
Description: IgG, IgM and IgA are disease related peripheral blood biomarkers used to assess disease progression of RA. A reduction in Ig values indicate an improvement in RA symptoms.
Time Frame: Baseline and Weeks 12, 24, 36, 52, and 72
Population: All enrolled participants with IgG, IgM or IgA assessment at 1 or more of the specified timepoints.
Measure: Mean (Standard Deviation); unit: Percent Change of Ig
Arm/Group | 120 mg LY2127399 Q4W
Number analyzed (Participants) | 26
Percent Change of Ig
  IgG Week 12 | -4.4 (13.0)
  IgG Week 24: number analyzed (Participants) | 24
  IgG Week 24 | -3.8 (11.0)
  IgG Week 36: number analyzed (Participants) | 23
  IgG Week 36 | -5.1 (12.1)
  IgG Week 52: number analyzed (Participants) | 21
  IgG Week 52 | -5.1 (14.2)
  IgG Week 72: number analyzed (Participants) | 19
  IgG Week 72 | -2.0 (14.5)
  IgM Week 12 | -7.7 (11.6)
  IgM Week 24: number analyzed (Participants) | 24
  IgM Week 24 | -9.3 (12.4)
  IgM Week 36: number analyzed (Participants) | 23
  IgM Week 36 | -11.6 (12.5)
  IgM Week 52: number analyzed (Participants) | 21
  IgM Week 52 | -12.4 (15.8)
  IgM Week 72: number analyzed (Participants) | 19
  IgM Week 72 | -9.0 (24.9)
  IgA Week 12 | -5.0 (12.9)
  IgA Week 24: number analyzed (Participants) | 24
  IgA Week 24 | -6.0 (14.5)
  IgA Week 36: number analyzed (Participants) | 23
  IgA Week 36 | -7.2 (15.4)
  IgA Week 52: number analyzed (Participants) | 21
  IgA Week 52 | -5.8 (13.2)
  IgA Week 72: number analyzed (Participants) | 19
  IgA Week 72 | -2.6 (20.1)

5. Secondary Outcome: Percent Change From Baseline in CD20+ B-cell Count
Description: CD20+ B-cells are a disease-related peripheral blood biomarker used to assess disease progression of RA. A reduction in CD20+ B-cell values indicate an improvement in RA symptoms.
Time Frame: Baseline and Weeks 12, 24, 36, 52, and 72
Population: All enrolled participants with CD20+ B-Cell assessment at 1 or more of the specified timepoints.
Measure: Mean (Standard Deviation); unit: Percent Change of cells
Arm/Group | 120 mg LY2127399 Q4W
Number analyzed (Participants) | 26
Percent Change of cells
  CD20+ B Week 12 | 3.8 (43.0)
  CD20+ B Week 24: number analyzed (Participants) | 24
  CD20+ B Week 24 | -17.3 (31.9)
  CD20+ B Week 36: number analyzed (Participants) | 22
  CD20+ B Week 36 | -20.8 (25.6)
  CD20+ B Week 52: number analyzed (Participants) | 21
  CD20+ B Week 52 | -32.0 (18.7)
  CD20+ B Week 72: number analyzed (Participants) | 19
  CD20+ B Week 72 | -44.6 (30.2)

6. Secondary Outcome: Percent Change From Baseline in Peripheral B-cell Subsets
Description: Peripheral B cell subsets (Mature Naive B-cells and Switched Memory B cells) are disease-related peripheral blood biomarkers used to assess disease progression of RA. A reduction in cell values indicate an improvement in RA symptoms.
Time Frame: Baseline and Weeks 12, 24, 36, 52, and 72
Population: All enrolled participants with Mature Naive B-Cells and Switched Memory B-Cells assessment at 1 or more of the specified timepoints.
Measure: Mean (Standard Deviation); unit: Percent Change of Cells
Arm/Group | 120 mg LY2127399 Q4W
Number analyzed (Participants) | 25
Percent Change of Cells
  Mature Naive B-Cell Week 12 | -10.8 (13.3)
  Mature Naive B-Cell Week 24: number analyzed (Participants) | 24
  Mature Naive B-Cell Week 24 | -14.9 (17.3)
  Mature Naive B-Cell Week 36: number analyzed (Participants) | 22
  Mature Naive B-Cell Week 36 | -18.2 (15.4)
  Mature Naive B-Cell Week 52: number analyzed (Participants) | 21
  Mature Naive B-Cell Week 52 | -19.6 (24.6)
  Mature Naive B-Cell Week 72: number analyzed (Participants) | 19
  Mature Naive B-Cell Week 72 | 7.6 (18.5)
  Switched Memory B-Cell Week 12 | 12.2 (54.6)
  Switched Memory B-Cell Week 24: number analyzed (Participants) | 24
  Switched Memory B-Cell Week 24 | 28.7 (76.7)
  Switched Memory B-Cell Week 36: number analyzed (Participants) | 22
  Switched Memory B-Cell Week 36 | 26.1 (57.3)
  Switched Memory B-Cell Week 52: number analyzed (Participants) | 21
  Switched Memory B-Cell Week 52 | 50.9 (106.8)
  Switched Memory B-Cell Week 72: number analyzed (Participants) | 19
  Switched Memory B-Cell Week 72 | 19.3 (61.2)

7. Secondary Outcome: Percent Change From Baseline in C-Reactive Protein (CRP)
Description: CRP is a disease-related peripheral blood biomarker used to assess disease progression of RA. A reduction in CRP values indicate an improvement in RA symptoms.
Time Frame: Baseline and Weeks 12, 24, 36, 52, and 72
Population: All enrolled participants with a CRP assessment at 1 or more of the specified timepoints.
Measure: Mean (Standard Deviation); unit: Percent Change of CRP
Arm/Group | 120 mg LY2127399 Q4W
Number analyzed (Participants) | 26
Percent Change of CRP
  CRP Week 12 | 63.0 (276.1)
  CRP Week 24: number analyzed (Participants) | 24
  CRP Week 24 | 15.4 (106.9)
  CRP Week 36: number analyzed (Participants) | 23
  CRP Week 36 | 19.0 (159.6)
  CRP Week 52: number analyzed (Participants) | 21
  CRP Week 52 | -4.9 (107.6)
  CRP Week 72: number analyzed (Participants) | 19
  CRP Week 72 | 7.1 (110.4)

8. Secondary Outcome: Percent Change From Baseline in Erythrocyte Sedimentation Rate (ESR)
Description: ESR is a disease related peripheral blood biomarker used to assess, in part, the effect of LY2127399 on the participants' RA disease progression. A reduction in ESR values indicate an improvement in RA symptoms.
Time Frame: Baseline and Weeks 12, 24, 36, 52, and 72
Population: All enrolled participants with an ESR assessment at 1 or more of the specific timepoints.
Measure: Mean (Standard Deviation); unit: Percent Change of ESR
Arm/Group | 120 mg LY2127399 Q4W
Number analyzed (Participants) | 26
Percent Change of ESR
  ESR Week 12: number analyzed (Participants) | 25
  ESR Week 12 | -4.2 (37.3)
  ESR Week 24: number analyzed (Participants) | 24
  ESR Week 24 | -7.8 (38.8)
  ESR Week 36: number analyzed (Participants) | 23
  ESR Week 36 | -7.3 (47.6)
  ESR Week 52: number analyzed (Participants) | 21
  ESR Week 52 | -4.0 (60.9)
  ESR Week 72: number analyzed (Participants) | 19
  ESR Week 72 | -5.0 (64.0)

ADVERSE EVENTS:
Groups:
- LY2127399 30 mg Q4W/120 mg Q4W: Participants who previously received 30 mg Q4W of LY2127399 in Study BCDK were assigned to receive120 mg of LY2127399 administered SC Q4W for 48 weeks.
- LY2127399 60 mg Q4W/120 mg Q4W: Participants who previously received 60 mg Q4W of LY2127399 in Study BCDK were assigned to receive120 mg of LY2127399 administered SC Q4W for 48 weeks.
- LY2127399 120 mg Q4W/120 mg Q4W: Participants who previously received 120 mg Q4W of LY2127399 in Study BCDK were assigned to receive120 mg of LY2127399 administered SC Q4W for 48 weeks.
- LY2127399 120 mg Q2W/120 mg Q4W: Participants who previously received 120 mg Q2W of LY2127399 in Study BCDK were assigned to receive120 mg of LY2127399 administered SC Q4W for 48 weeks.
Arm/Group | Placebo/LY2127399 120 mg Q4W | LY2127399 30 mg Q4W/120 mg Q4W | LY2127399 60 mg Q4W/120 mg Q4W | LY2127399 120 mg Q4W/120 mg Q4W | LY2127399 120 mg Q2W/120 mg Q4W
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/6 | 0/4 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 5/6 | 4/6 | 4/4 | 3/5 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo/LY2127399 120 mg Q4W (N=6) | LY2127399 30 mg Q4W/120 mg Q4W (N=6) | LY2127399 60 mg Q4W/120 mg Q4W (N=4) | LY2127399 120 mg Q4W/120 mg Q4W (N=5) | LY2127399 120 mg Q2W/120 mg Q4W (N=5)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo/LY2127399 120 mg Q4W (N=6) | LY2127399 30 mg Q4W/120 mg Q4W (N=6) | LY2127399 60 mg Q4W/120 mg Q4W (N=4) | LY2127399 120 mg Q4W/120 mg Q4W (N=5) | LY2127399 120 mg Q2W/120 mg Q4W (N=5)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Keratoconjunctivitis sicca (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enteritis infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Mycoplasma infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 3 (4)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transfusion (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days